CLINICAL TRIAL: NCT06668129
Title: Effects of a Postural Education Multicomponent Intervention in Primary School Children.
Acronym: PEPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: State Research Agency, Spain (Other Government); European Regional Development Fund (Other); Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 130CER19; RTI2018-101023-A-I00 (Other Grant/Funding Number: Spanish Ministry of Science, Innovation and Universities)
Record Dates: First submitted 2024-10-21; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Physical Activity; Back Pain Lower Back
MeSH Terms: conditions — Motor Activity; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back care intervention program (Experimental)
  Interventions: Behavioral: Back care intervention program
- Control condition (No Intervention)

INTERVENTIONS:
Behavioral: Back care intervention program — The back care intervention consists of:
  1. Nine oral presentations. Include "Programa Suma't" programme developed by the Provincial Council of Majorca.
  2. Multisubject Teaching Unit.
  3. Information campaign widespread by the school (i.e. posters, triptychs, school website, social networks, etc.)
  4. "The Back Care Day" at school.
  Arms: Back care intervention program

SUMMARY:
The present study, named PEPE project, aims to study the effects of a 9-month postural educational multicomponent intervention on back health in schoolchildren. As well as, this project aims to examine the effectiveness of the intervention on teachers. Total of 2000 children aged 10 to 12 and 20 schools will be randomized into an intervention group (N=1000 children, N=10 schools) and a control group (N=1000 children, N=10 schools). A 9-months intervention program will be implemented. Participants will be evaluated three times: before the intervention (baseline, Month 0), after the intervention (post-test, Month 9) and 6 months after the intervention finished (follow-up, Month 15). The intervention will consist on: (1) nine oral presentations delivered at school, (2) multisubject teaching unit, (3) information campaign widespread by the school (i.e. posters, triptychs, school website, social networks, etc.), and (4) The Back-Care Day at school. The effectiveness of the intervention will be evaluated by means of primary outcomes which include the back-care knowledge of schoolchildren. As well as, a set of secondary outcomes such as daily postural habits, use of a backpack, and LBP prevalence in schoolchildren and among teachers involved will be studied. This intervention will provide new insights into the prevention of childhood LBP which may lead to a better management of this health problem throughout an individuals lifetime.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 10 and 12 years, who belonged to the fifth and sixth grades of primary school.

Exclusion Criteria:

* Children with some type of medical condition that may affect the results of the measurements or that present some limitation of their abilities that prevents the intervention program from developing normally.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 849 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Knowledge of back health | 16 weeks
  Validated questionnaire with Spanish children (Cronbach's alpha = 0.82) will be used to ascertain children's' level of knowledge on back care in daily life physical activities. Specifically, this questionnaire has 24 multiple choice items associated with one of the following categories according to conceptual knowledge: topographicalanatomical knowledge (items 1, 2, 3 and 6); functional-anatomical knowledge (items 4, 5 and 7); habits in standing posture (items 8-10); or seated (items 11-13); or lying (items 23 and 24); habits in carrying heavy objects in a backpack (items 14-18); and how to move heavy loads (items 19-22).
  Additionally, the questionnaire validated with Spanish schoolchildren and used in Méndez et al. will be used to assess back posture knowledge related to general principles of good body mechanics and fear-avoiding beliefs.

SECONDARY OUTCOMES:
Daily postural habits | 16 weeks
  Daily life habits will be assessed by means of a questionnaire that will be fulfilled by the children. The questionnaire include the following items: being allowed to leave the academic material at school (yes=1/no=0), correct use of sofa (yes/no), stooping correctly (yes/no), take care to sit correctly at home (yes/no), take care to sit correctly at school (yes/no), frequent posture change on chair at home (yes/no), and frequent posture change on chair at school (yes/no).
Backpack use | 16 weeks
  Correct use of backpack will be assessed by means of a questionnaire that will be fulfilled by the children. The questionnaire include the following items: try to load the minimum weight possible, carry a backpack on two shoulders, belief that school backpack weight does not affect the back and the use of a locker or similar at school.
  The weight of the children's' backpack will be also measured.
LBP prevalence | 16 weeks
  The instrument to evaluate LBP prevalence will be based using a validated questionnaire. Data related to LBP included in the questionnaire were the following: LBP experience during the student's lifetime (never, almost never, sometimes, often, always), LBP impeding usual activities (never, only when in pain, always), treatment received for LBP (no, rehabilitation, drugs, surgery, others), LBP in bed during the night or upon waking (yes, no), LBP during the last week (yes, no), LBP during or at the end of a physical education (PE) class (never, almost never, sometimes, often, always), diagnosis of scoliosis and diagnosis of different leg length (yes, no).
Back care knowledge | 16 weeks
  Low Back Pain Knowledge Questionnaire (LKQ) will be used as an instrument to assess knowledge about back pain in teachers. This questionnaire is composed of 16 questions, divided into the following categories: general aspects, concepts, and treatment. The total maximum score is 24 and is classified into one of three levels: low (0 - 14), moderate (15 - 18), and high (19 - 24).
LBP prevalence and daily postural habits | 16 weeks
  The Quebec Back Pain Disability Scale will be used to assess daily postural habits of teachers. The scale exists of one central question: "Do you have trouble today with...?" followed by 20 activities of daily life. In every activity, there are 6 answer categories, measured by using a Likert scale from 0-5 (0 = no effort, 5 = not able to). The final outcome is obtained by the sum of the scoring of the degree of difficulty in performing the 20 daily activities. These outcomes score within the range of 0 and 100, determents the level of functional disability, with higher numbers representing greater levels of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Balearic Islands, Palma, Balearic Islands, Spain